CLINICAL TRIAL: NCT04084704
Title: A Prospective Evaluation of the Cingal Injection for Hip Osteoarthritis (ECHO Study)
Brief Title: A Prospective Evaluation of the Cingal Injection for Hip Osteoarthritis
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Anika Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Olufemi Ayeni, Principal Investigator, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7692
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cingal injection (Other): Cingal will be administered by fellowship-trained physicians through ultrasound-guided injection using a 21-gauge needle into the joint space of the hip under sterile conditions. The needle track will be anesthetized with local anesthetic.
  Interventions: Device: Cingal

INTERVENTIONS:
Device: Cingal — Cingal will be administered by fellowship-trained physicians through ultrasound-guided injection using a 21-gauge needle into the joint space of the hip under sterile conditions. The needle track will be anesthetized with local anesthetic.

SUMMARY:
Osteoarthritis (OA) of the hip is one of the ten most disabling diseases in the developed world. Because OA gradually worsens over time, the sooner treatment is started, the more likely its impact is lessened. Hip OA is characterized by joint pain, cartilage degeneration, and an increase in disability. Multiple treatments are used to manage the degenerating hip as well as the associated pain. These include physiotherapy and rehabilitation, bracing, other walking aids, oral medications, injections, and in severe cases, surgery. Prior research has shown that injection of hyaluronic acid (HA) and corticosteroids can slow down OA degradation. This study will look at the effects of injecting Cingal into the hip, which expands on its current approved use in the treatment of knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women ages 40 to 65 years
2. Hip OA (mild to moderate) diagnosed on x-ray and/or MRI (Tonnis grade 1 and 2)
3. Patient is using only nonsteroidal anti-inflammatory drugs (NSAIDs) or acetaminophen/ paracetamol (Tylenol) for pain relief during the month before receiving Cingal
4. Patient is willing to stop pain/anti-inflammatory medication at least two weeks prior to receiving Cingal through the end of the study (6 months)
5. Patient speaks, reads, and understands the language of the clinical site
6. Provision of informed consent

Exclusion Criteria:

1. Evidence of hip dysplasia (centre edge angle less than 20 degrees)
2. Presence of advanced hip OA (Tonnis Grade 3)
3. Previous trauma to the affected hip requiring medical or surgical treatment
4. Previous surgery on the affected hip or contralateral hip
5. Severe acetabular deformities (e.g. acetabular protrusion, coxa profunda, circumferential labral ossification)
6. Infections or skin diseases at target hip joint
7. Immunosuppressive medication use
8. Chronic pain syndromes
9. Significant medical co-morbidities (requiring daily assistance for activities of daily living)
10. History of paediatric hip disease (e.g. Legg-Calve-Perthes; slipped capital femoral epiphysis)
11. Previous cartilage repair procedure (microfracture, Osteochondral Autograft Transplantation System (OATS) or Autologous Chondrocyte Implantation (ACI) with or without use of a scaffold (matrix) in the index hip)
12. Known hypersensitivity (allergy) to hyaluronan preparations
13. Known hypersensitivity (allergy) to triamcinolone hexacetonide preparations
14. Known sensitivity to any of the materials in Cingal
15. Patients with impaired cardio-renal function, endocrine, or other diseases or conditions that use of corticosteroid is warned
16. HA intra-articular injections into the index hip within the last 6 months before receiving Cingal
17. Corticosteroid therapy by systemic, intra-articular, or intramuscular route or oral corticosteroids within the last 6 months before receiving Cingal
18. Any injection received in the hip prior to receiving or received concurrently with Cingal
19. Uncontrolled diabetes
20. Subject is a woman who is pregnant or breastfeeding or a woman of child bearing potential who refuses to use effective contraception during the course of the study
21. Patient is incarcerated
22. Any clinically significant or symptomatic vascular or neurologic disorder of the lower extremities
23. Rheumatoid arthritis or gouty arthritis
24. Current diagnosis of osteomyelitis
25. Diagnosed musculoskeletal cancer or any diagnosed cancer, other than musculoskeletal if not on long term remission (e.g. at least 5 years or negative biopsy at last exam), except basal cell carcinoma
26. Patients who are at higher risk for post-surgical bleeding (e.g., bleeding disorder; taking anticoagulants except low dose aspirin or anti-platelet agents [e.g. ASA, Plavix]) or post-surgical infection (e.g., taking immunosuppressants; have a severe infection or a history of serious infection)
27. Participation in concurrent trial that involves a medical intervention
28. Patient is currently receiving workman's compensation or disability, has been involved in an motor vehicle accident, or is in litigation for workman's compensation or disability claims
29. Likely problems, in the judgment of the treating physician, with maintaining follow up (e.g. patients with no fixed address, plans to move out of town). This may include patients with severe mental disorders and drug addictions without adequate support.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Patient reported hip pain as measured by Visual Analog Scale | 6 months
  The primary objective of this observational study is to determine, among individuals with hip OA ages 40-65 years, the effect of Cingal on patient-reported hip pain, as measured by a Visual Analogue Scale (VAS), at 6-months post-injection.

SECONDARY OUTCOMES:
Hip Function, as measured by the Hip Disability and Osteoarthritis Outcome Score (HOOS) | 6 months
  The HOOS was designed to assess patient opinions about their hip and associated problems in an adult population with a hip disability with or without OA. The HOOS has been extensively validated and consists of 5 subscales for pain, other symptoms, function in activities of daily living, function in sports and recreation, and hip-related quality of life.
Health-related quality of life (HRQL) as measured by the Short Form-12 questionnaire (SF-12) | 6 months
  The SF-12 may be self or interview-administered and can help document mental and physical components of quality of life. Points can range from 0-100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health.
Physical activity levels as measured by a wrist-worn activity tracker | 6 months
  To be worn for one week prior to each follow-up visit.
Complications, including infection and other adverse events at 6-months post-injection. | 6 months
  Adverse events
Range of motion | 6 months
  ROM will be measured with standard anterior and posterior impingement tests, the log roll test, and hip flexion/extension, abduction/adduction, and internal/external rotation.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No